CLINICAL TRIAL: NCT02207660
Title: Cisplatin Plus One Day 24 Hour Infusion of High-Dose 5-Fluorouracil for Stage IVB, Recurrent or Metastatic Carcinoma of the Uterine Cervix.
Brief Title: Cisplatin Plus One-Day 24-hour Infusion of High-Dose 5-Fluorouracil for Stage IVB, Recurrent or Metastatic Carcinoma of the Uterine Cervix
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201211032RIC
Record Dates: First submitted 2013-07-03; First posted 2014-08-04 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Cervical Cancer
Keywords: cisplatin; Cervical cancer; metastasis; recurrence
MeSH Terms: conditions — Uterine Cervical Neoplasms; Neoplasm Metastasis; Recurrence | interventions — Fluorouracil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cisplatin,P-HDFL: The general principles for patients schedule for P-HDFL regimen treatment were as followings: patients must have had white cell count > 3000/mm3, platelet count > 100000/mm3, a normal serum creatinine (≦1.5 mg/dL) or a measured creatinine clearance ([urine creatinine level (mg/dL) X 24-hr urine amount (mL)]/[serum creatinine level (mg/dL) X 1,440 min]) of ≧ 40 mL/min [12,15], total bilirubin ≦ 2 mg/dL, and transaminase (≦3X the upper normal limits). Also, patients needed to have measurable disease by radiographic studies (plain X-ray, CT or MRI scans), no serious active underlying medical issues, and Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
  Interventions: Drug: Cisplatin,P-HDFL

INTERVENTIONS:
Drug: Cisplatin,P-HDFL — The P-HDFL regimen was given as follows: In each 21-day cycle, patients received 24-hour infusions of cisplatin at 45 or 50 mg/m2 and 5-FU 2,600mg/m2 plus leucovorin 300 mg/m2 intravenous 24-hour infusion on Day 1. Normal saline hydration (≧1000 mL), dexamethasone, and antiemetics (ondansetron or granisetron) were given prophylactically before each dose of cisplatin.
  Other Names: Abilatin、Platamine、Platinex; fluorouracil

SUMMARY:
Objectives: To evaluate the effectiveness and toxicity of the combination of infusional cisplatin and 24-hour infusion of high-dose fluorouracil plus leucovorin (P-HDFL) repeatedly every 21 days for the treatment of stage IVB, recurrent or metastatic carcinoma of cervix.

Methods: The medical records of all patients with stage IVB, recurrent or metastatic cervical cancer who were treated with P-HDFL regimen between January 2005 and December 2009 at National Taiwan University Hospital were reviewed.

Expected results: Investigators will identify the effectiveness and toxicity of the combination of infusional cisplatin and 24-hour infusion of high-dose fluorouracil plus leucovorin (P-HDFL) repeatedly every 21days for the treatment of stage IVB, recurrent or metastatic carcinoma of cervix.

DETAILED DESCRIPTION:
The medical records for all patients with advanced, metastatic or recurrent cervical cancer who were treated with P-HDFL regimen between January 2005 and December 2009 at National Taiwan University Hospital were reviewed. Recurrences were confirmed by histopathologic examinations. Cases of recurrent cervical cancer, who undergoing salvage surgery and receiving P-HDFL as adjuvant therapy, were excluded from this study. The general principles for patients schedule for P-HDFL regimen treatment were as followings: patients must have had white cell count > 3000/mm3, platelet count > 100000/mm3, a normal serum creatinine (≦1.5 mg/dL) or a measured creatinine clearance ([urine creatinine level (mg/dL) X 24-hr urine amount (mL)]/[serum creatinine level (mg/dL) X 1,440 min]) of ≧ 40 mL/min [12,15], total bilirubin ≦ 2 mg/dL, and transaminase (≦3X the upper normal limits). Also, patients needed to have measurable disease by radiographic studies (plain X-ray, CT or MRI scans), no serious active underlying medical issues, and Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2. The ethical approval for this retrospective study was obtained from our research ethics committee in this hospital.

The P-HDFL regimen was given as follows: In each 21-day cycle, patients received 24-hour infusions of cisplatin at 45 or 50 mg/m2 and 5-FU 2,600mg/m2 plus leucovorin 300 mg/m2 intravenous 24-hour infusion on Day 1. Normal saline hydration (≧1000 mL), dexamethasone, and antiemetics (ondansetron or granisetron) were given prophylactically before each dose of cisplatin.

Physical examination, survey of adverse reactions and hemogram checkup of patients were performed before administering each dose of the P-HDFL treatment. Tumor response and toxicity were evaluated according to the World Health Organization criteria [16]. A complete response (CR) was defined as the disappearance of all measurable disease for at least 4 weeks. A partial response (PR) was defined as a 50% or more reduction in the products of each measurable lesion for at least 4 weeks. Progressive disease (PD) was defined as a 25% or more increase in the size of one or more measurable lesions or the appearance of new lesions. Stable disease (SD) was defined as any condition not meeting any the above criteria.

Progression-free survival was measured from the first date of chemotherapy to the date of documented disease progression, death of other causes or last contact. Overall survival was measured from the first date of chemotherapy to death or last contact. Progression-free survival and overall survival were estimated by using the method of Kaplan-Meier.

ELIGIBILITY:
Inclusion Criteria:

* all patients with stage IVB, recurrent or metastatic cervical cancer who were treated with P-HDFL

Exclusion Criteria:

* Cases of recurrent cervical cancer, who undergoing salvage surgery and receiving P-HDFL as adjuvant therapy, were excluded from this study.

Ages: 20 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The general principles for patients schedule for P-HDFL regimen treatment were as followings: patients must have had white cell count > 3000/mm3, platelet count > 100000/mm3, a normal serum creatinine (≦1.5 mg/dL) or a measured creatinine clearance ([urine creatinine level (mg/dL) X 24-hr urine amount (mL)]/[sereum creatinine level (mg/dL) X 1,440 min]) of ≧ 40 mL/min [12,15], total bilirubin ≦ 2 mg/dL, and transaminase (≦3X the upper normal limits). Also, patients needed to have measurable disease by radiographic studies (plain X-ray, CT or MRI scans), no serious active underlying medical issues, and Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-07; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | 5 years
  From the first date of chemotherapy to death or last contact.

SECONDARY OUTCOMES:
Progression-free survival | 5 years
  From the first date of chemotherapy to the date of documented disease progression, death of other causes or last contact.

CONTACTS AND LOCATIONS:
Overall Officials: Chi-An Chen, MD, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan